CLINICAL TRIAL: NCT02480361
Title: Effect of Acupuncture on Postoperative Ileus After Gastrectomy in Patients With Gastric Cancer: A Pilot Study
Brief Title: Effect of Acupuncture on Postoperative Ileus After Gastric Surgery (EAPIG)
Acronym: EAPIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, In-Hwan Kim, Doctor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APOIGC-13
Record Dates: First submitted 2015-06-09; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Ileus
Keywords: Acupuncture; Gastric cancer
MeSH Terms: conditions — Ileus; Stomach Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): The patients who were received acupuncture after gastric cancer surgery
  Interventions: Device: acupuncture
- Non-acupuncture (No Intervention): The patients who were not received acupuncture after gastric cancer surgery

INTERVENTIONS:
Device: acupuncture — Acupuncture treatment after gastric cancer surgery during 5 postoperative days
  Arms: Acupuncture

SUMMARY:
Postoperative ileus (POI) is a common problem after major abdominal surgery. Acupuncture is being accepted in the West as a treatment option for managing POI and various functional gastrointestinal disorders. Therefore, we conducted a prospective randomized pilot study to evaluate the effect of electro-acupuncture on POI and other surgical outcomes in patients who underwent gastric surgery for a later large-scale study.

DETAILED DESCRIPTION:
Before surgery, patients were randomized (using simple randomization) to either acupuncture (A) group or non-acupuncture (NA) group. In both groups, sitz markers were inserted in duodenum or jejunum during surgery for detection of postoperative remnant sitz markers by Xray. In the A group, acupuncture treatment was given once daily for up to 5 consecutive days starting on postoperative day 1. The acupuncture points which were used were based on traditional Korean medicine. No acupuncture treatment was performed in the NA group.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery for gastric cancers
* Patients with American Society of Anesthesiologists grades I-III
* Patients who provided written informed consent

Exclusion Criteria:

* Patients who developed intraoperative problems or complications
* Patients with contraindications to had electrical stimulation devices (pacemaker or implantable defibrillator)
* Patients who were allergic to acupuncture needle

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Remnant sitz markers in small intestine at postoperative day 1 | measured in postoperative day 1
  Numbers of of remnant sitz markers in the small intestine that did not pass through ileo-cecal valve, measured by X-ray on postoperative day 1.
Remnant sitz markers in small intestine at postoperative day 3 | measured in postoperative day 3
  Numbers of of remnant sitz markers in the small intestine that did not pass through ileo-cecal valve, measured by X-ray on postoperative day 3.
Remnant sitz markers in small intestine at postoperative day 5 | measured in postoperative day 5
  Numbers of of remnant sitz markers in the small intestine that did not pass through ileo-cecal valve, measured by X-ray on postoperative day 5.
Remnant sitz markers in small intestine at postoperative day 7 | measured in postoperative day 7
  Numbers of of remnant sitz markers in the small intestine that did not pass through ileo-cecal valve, measured by X-ray on postoperative day 7.

SECONDARY OUTCOMES:
Time to first flatus | up to 5 dyas
start of water intake | up to 7days
start of soft diet | up to 7days
hospital stay | up to 2 weeks

OTHER OUTCOMES:
white blood cell count in preoperative period | measured in day before operation
white blood cell count in postoperative day 1 | measured in postoperative day 1
white blood cell count in postoperative day 3 | measured in postoperative day 3
white blood cell count in postoperative day 5 | measured in postoperative day 5
white blood cell count in postoperative day 7 | measured in postoperative day 7
serum C reactive protein level in preoperative period | measured in day before operation
serum C reactive protein level in postoperative day 1 | measured in postoperative day 1
serum C reactive protein level in postoperative day 3 | measured in postoperative day 3
serum C reactive protein level in postoperative day 5 | measured in postoperative day 5
serum C reactive protein level in postoperative day 7 | measured in postoperative day 7
serum albumin level in preoperative period | measured in day before operation
serum albumin level in postoperative day 1 | measured in postoperative day 1
serum albumin level in postoperative day 3 | measured in postoperative day 3
serum albumin level in postoperative day 5 | measured in postoperative day 5
serum albumin level in postoperative day 7 | measured in postoperative day 7

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-dong Chae, Professor, Study Director — Department of Surgery, School of Medicine, Catholic University of Daegu